CLINICAL TRIAL: NCT02678312
Title: Multicenter, Open-label Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LCZ696 Followed by a 52-week Randomized, Double-blind, Parallel Group, Active-controlled Study to Evaluate the Efficacy and Safety of LCZ696 Compared With Enalapril in Pediatric Patients From 1 Month to < 18 Years of Age With Heart Failure Due to Systemic Left Ventricle Systolic Dysfunction
Brief Title: Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of LCZ696 Followed by a 52-week, Double-blind Study of LCZ696 Compared With Enalapril in Pediatric Patients With Heart Failure
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLCZ696B2319; 2015-004207-22 (EudraCT Number)
Record Dates: First submitted 2016-02-04; First posted 2016-02-09 (Estimated); Results first posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-01

CONDITIONS: Pediatric Heart Failure
Keywords: Pediatric Heart failure,; systemic left ventricle,; reduced ejection fraction
MeSH Terms: interventions — sacubitril and valsartan sodium hydrate drug combination; Enalapril

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (3):
- Part 1: LCZ696 open label (Experimental): LCZ696 open label: For Age Groups 1 and 2, either 1) 0.8 mg/kg or 2) 3.1 mg/kg or both. For Age Group 3, either 1) 0.4 mg/kg or 2) 1.6 mg/kg or both. After LCZ696 PK assessment, patients will be maintained on open-label Enalapril provided locally by the study site, or standard of care also provided locally by the study site, for heart failure treatment, if patient intended to participate in Part 2.
  Interventions: Drug: LCZ696; Drug: Enalapril
- Part 2: Enalapril (Active Comparator): The target dose for enalapril is 0.2 mg/kg bid (0.4 mg/kg total daily dose) with a maximum dose of 10 mg bid (20 mg total daily dose). Administered in a double-blind fashion.
  Interventions: Drug: Enalapril; Drug: Placebo of LCZ696
- Part 2: LCZ696 (Experimental): LCZ696 3.125 mg granules and adult formulation (50, 100, 200 mg) can be given based on patient weight. Administered in a double-blind fashion.
  Interventions: Drug: LCZ696; Drug: Placebo of Enalapril

INTERVENTIONS:
Drug: LCZ696 — LCZ696: 3.125 mg granules (packaged in capsules containing 4 or 10 granules)
  Arms: Part 1: LCZ696 open label; Part 2: LCZ696
Drug: Enalapril — Enalapril tablets: 2.5 mg, 5 mg, 10 mg dosage strengths
  Arms: Part 1: LCZ696 open label; Part 2: Enalapril
Drug: Placebo of LCZ696
  Arms: Part 2: Enalapril
Drug: Placebo of Enalapril
  Arms: Part 2: LCZ696
Drug: LCZ696 — LCZ696: 3.125 mg granules (packaged in capsules containing 4 or 10 granules), tablets: 50 mg, 100 mg, 200 mg dosage strengths
  Arms: Part 2: LCZ696

SUMMARY:
This study consists of two parts (Part 1 and Part 2). The purpose of Part 1 is to evaluate the way the body absorbs, distributes, metabolizes and removes the drug LCZ696. This will help determine the proper dose of LCZ696 for Part 2 of the study.

The purpose for Part 2 is to compare the effectiveness and safety of LCZ696 with enalapril in a double-blind manner, in pediatric heart failure patients over 52 weeks of treatment.

DETAILED DESCRIPTION:
This study consists of two parts (Part 1 and Part 2). The purpose of Part 1 is to evaluate the way the body absorbs, distributes, metabolizes and removes the drug LCZ696. This will help determine the proper dose of LCZ696 for Part 2 of the study.

The purpose for Part 2 is to compare the effectiveness and safety of LCZ696 with enalapril in a double-blind manner, in pediatric heart failure patients over 52 weeks of treatment.

ELIGIBILITY:
Key Inclusion Criteria:

* Chronic heart failure (CHF) resulting from left ventricular systolic dysfunction, and receiving chronic HF therapy (if not newly diagnosed)
* New York Heart Association (NYHA) classification II-IV (older children: 6 to <18 years old) or Ross CHF classification II-IV (younger children: < 6 years old)
* Systemic left ventricular ejection fraction ≤ 45% or fractional shortening ≤22.5%
* For Part 1 study: Patients must be treated with an angiotensin converting enzyme inhibitor (ACEI) or angiotensin receptor blockers (ARB) prior to screening. Patients in Group 1 and 2 must be currently treated with the dose equivalent of at least enalapril 0.2 mg/kg prior to the LCZ696 3.1 mg/kg administration. Group 3 patients will participate in LCZ696 0.8 mg/kg and not LCZ696 3.1 mg/kg.
* Biventricular physiology with systemic left ventricle

Key Exclusion Criteria:

* Patient with single ventricle or systemic right ventricle
* Patients listed for heart transplantation (as United Network for Organ Sharing status 1A) or hospitalized waiting for transplant (while on inotropes or with ventricular assist device)
* Sustained or symptomatic dysrhythmias uncontrolled with drug or device therapy
* Patients that have had cardiovascular surgery or percutaneous intervention to palliate or correct congenital cardiovascular malformations within 3 months of the screening visit. Patients anticipated to undergo corrective heart surgery during the 12 months after entry into Part 2
* Patients with unoperated obstructive or severe regurgitant valvular (aortic, pulmonary, or tricuspid) disease, or significant systemic ventricular outflow obstruction or aortic arch obstruction
* Patients with restrictive or hypertrophic cardiomyopathy
* Active myocarditis
* Renal vascular hypertension (including renal artery stenosis)
* Moderate-to severe obstructive pulmonary disease
* Serum potassium > 5.3 mmol/L
* History of angioedema
* Allergy or hypersensitivity to ACEI / ARB

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 393 (Actual)
Dates: Start 2016-11-03 (Actual); Primary Completion 2022-01-03 (Actual); Study Completion 2022-01-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (90):
- United States (23):
  - Novartis Investigative Site, Loma Linda, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Palo Alto, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Aurora, Colorado
  - Novartis Investigative Site, Gainesville, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, St. Petersburg, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Ann Arbor, Michigan
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Rochester, Minnesota
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Salt Lake City, Utah
  - Novartis Investigative Site, Seattle, Washington
- Argentina (2):
  - Novartis Investigative Site, Ramos Mejía, Buenos Aires
  - Novartis Investigative Site, Salta, Salta Province
- Novartis Investigative Site, Innsbruck, Austria
- Novartis Investigative Site, Sofia, Bulgaria
- Canada (2):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Toronto, Ontario
- China (3):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
- Novartis Investigative Site, Zagreb, Croatia
- Novartis Investigative Site, Prague, Czechia
- Novartis Investigative Site, Helsinki, Finland
- France (3):
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pessac
- Germany (6):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Stuttgart
- Novartis Investigative Site, Budapest, Hungary
- India (3):
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Kochi, Kerala
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
- Novartis Investigative Site, Beersheba, Israel
- Italy (8):
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Napoli
- Japan (8):
  - Novartis Investigative Site, Ōbu, Aichi-ken
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Ōmura, Nagasaki
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Setagaya-ku, Tokyo
  - Novartis Investigative Site, Shinjuku Ku, Tokyo
  - Novartis Investigative Site, Toyama, Toyama
  - Novartis Investigative Site, Saitama
- Novartis Investigative Site, Amman, JOR, Jordan
- Lebanon (2):
  - Novartis Investigative Site, Beirut
  - Novartis Investigative Site, El Achrafîyé
- Poland (2):
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Warsaw
- Portugal (3):
  - Novartis Investigative Site, Carnaxide, Lisbon District
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Lisbon
- Russia (2):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- Novartis Investigative Site, Riyadh, Saudi Arabia
- Novartis Investigative Site, Singapore, Singapore
- South Korea (2):
  - Novartis Investigative Site, Yangsan, Gyeongsangnam-do
  - Novartis Investigative Site, Seoul
- Spain (3):
  - Novartis Investigative Site, Córdoba, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Lausanne, Switzerland
- Taiwan (2):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taipei
- Thailand (2):
  - Novartis Investigative Site, Bangkoknoi, Bangkok
  - Novartis Investigative Site, Bangkok
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Konak

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel based on scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Shaddy R, Burch M, Kantor PF, Solar-Yohay S, Garito T, Zhang S, Kocun M, Mao C, Cilliers A, Wang X, Canter C, Rossano J, Wallis G, Menteer J, Daou L, Kusa J, Tokel K, Dilber D, Xu Z, Xiao T, Halnon N, Daly KP, Bock MJ, Zuckerman W, Singh TP, Chakrabarti M, Levitas A, Senni M, Grutter G, Kim GB, Song J, Lee HD, Chen CK, Sanchez-de-Toledo J, Law Y, Wanitkun S, Cui Y, Anjos R, Mese T, Bonnet D; PANORAMA-HF Investigators. Sacubitril/Valsartan in Pediatric Heart Failure (PANORAMA-HF): A Randomized, Multicenter, Double-Blind Trial. Circulation. 2024 Nov 26;150(22):1756-1766. doi: 10.1161/CIRCULATIONAHA.123.066605. Epub 2024 Sep 25. PMID 39319469
- [Derived] Shaddy R, Burch M, Kantor PF, Solar-Yohay S, Garito T, Zhang S, Kocun M, Bonnet D. Baseline Characteristics of Pediatric Patients With Heart Failure Due to Systemic Left Ventricular Systolic Dysfunction in the PANORAMA-HF Trial. Circ Heart Fail. 2023 Mar;16(3):e009816. doi: 10.1161/CIRCHEARTFAILURE.122.009816. Epub 2023 Jan 5. PMID 36601956

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2-Part (Pt) Study: Pt 1 a single dose PK/PD study with 2 dose levels; Pt 2 is a 52-week, double blind, active controlled, randomized, safety & efficacy study. In Pt 1, there were 3 age groups: 6 to <18 yrs, 1 to <6 yrs and 1 month to <1 yr. Each received either a single low dose LCZ696 (Cohort 1), a single high dose LCZ696 (Cohort 2) or both. Cohort S included patients receiving a single low dose after having received a single high dose. The low/high doses for groups 1/2 were 0.8 & 3.1 (mg/kg).
Pre-assignment Details: The low and high doses for Group 3 0.4 mg/kg and 1.6 mg/kg, respectively. 26 patients received either one or two single doses of LCZ696 in Pt 1. In Pt 2, patients were randomized to receive either LCZ696 or enalapril. 377 patients were randomized and 375 received study drug (2 did not receive drug). 11 of 26 Pt 1 patients rolled into Pt 2; however, 1 patient had two ID numbers; so only 10 unique patients were in Pt 1 & 2.
Groups:
- Part 1: Dose Cohort 1: Participants received LCZ696 0.4 mg/kg (age group 3 {1 month to < 1 year}) or 0.8 mg/kg (age group 1 {6 to <18 years} and age group 2 {1 to < 6 years}), based on age, given as a single oral dose on Day 1 of period 1.
- Part 1: Dose Cohort 2: Participants received LCZ696 1.6 mg/kg (age group 3 {1 month to < 1 year}) or 3.1 mg/kg (age group 1 {6 to <18 years} and age group 2 {1 to < 6 years}), based on age, given as a single oral dose on Day 1 of period 2.
- Part 1: Dose Cohort S: Participants in the dose cohort 2 who received LCZ696 3.1 mg/kg on Day 1 of period 2 and later received LCZ696 0.8 mg/kg, within period 2.
- Part 2: LCZ696: Participants received LCZ696 3.1 mg/kg (age group 1 {6 to <18 years} and age group 2 {1 to < 6 years}) or 2.3 mg/kg (age group 3 {1 month to < 1 year}), based on age, orally, twice a day (BID) for 52 weeks.
- Part 2: Enalapril: Participants received enalapril 0.2 mg/kg (age group 1 {6 to <18 years} and age group 2 {1 to < 6 years}) or 0.15 mg/kg (age group 3 {1 month to < 1 year}), based on age, orally, BID, for 52 weeks.
Period: Part 1 Open Label Epoch- Period 1
Arm/Group | Part 1: Dose Cohort 1 | Part 1: Dose Cohort 2 | Part 1: Dose Cohort S | Part 2: LCZ696 | Part 2: Enalapril
Started (Out of 26 participants enrolled in the Part 1 of the study, 17 were dosed based on their age to receive LCZ696 0.8 mg or 0.4 mg in Period 1.) | 17 | 0 | 0 | 0 | 0
Completed | 14 | 0 | 0 | 0 | 0
Not Completed | 3 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0
Period: Part 1 Open Label Epoch- Period 2
Arm/Group | Part 1: Dose Cohort 1 | Part 1: Dose Cohort 2 | Part 1: Dose Cohort S | Part 2: LCZ696 | Part 2: Enalapril
Started | 0 | 18 (Out of 26 participants enrolled in Part 1, 18 participants were dosed in dose cohort 2 to receive LCZ696 1.6 mg or 3.1 mg dose in Period 2. A total of 9 participants who received LCZ696 in Dose cohort 1, received drug further in dose cohort 2 and 9 others received drug directly in Period 2 were included in Dose cohort 2.) | 2 (2 participants who were dosed in Dose Cohort 2 at dose level 3.1 mg/kg were then prescribed one dose of study drug at dose level 0.8 mg/kg within period 2 and were therefore grouped under Dose cohort S.) | 0 | 0
Completed | 0 | 18 | 2 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Part 2 Double Blind Epoch
Arm/Group | Part 1: Dose Cohort 1 | Part 1: Dose Cohort 2 | Part 1: Dose Cohort S | Part 2: LCZ696 | Part 2: Enalapril
Started (Out of 377 participants enrolled in Part 2 of the study, 2 participants in the enalapril arm were randomized in error and did not receive the study medication. Therefore, 375 of 377 randomized participants received study medication.) | 0 | 0 | 0 | 187 | 188
Completed | 0 | 0 | 0 | 169 | 164
Not Completed | 0 | 0 | 0 | 18 | 24
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 2
Not completed — Death | 0 | 0 | 0 | 8 | 12
Not completed — Technical Problems | 0 | 0 | 0 | 4 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 2
Not completed — Subject/guardian Decision | 0 | 0 | 0 | 5 | 6

BASELINE CHARACTERISTICS:
Population: Full Analysis Set included all randomized participants who received study drug, with the exception of [2 patients in Part 2] who had not received any study drug, but had been inadvertently randomized into the study (mis-randomized).
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Dose Cohort 1 | Part 1: Dose Cohort 2 | Part 1: Dose Cohort S | Part 2: LCZ696 | Part 2: Enalapril | Total
Number analyzed (Participants) | 17 | 18 | 2 | 187 | 188 | 412
Age, Continuous [Median (Full Range); unit: years] | 3.00 [0.30 to 16.00] | 2.50 [0.20 to 17.00] | 1.55 [1.10 to 2.00] | 7.00 [0.50 to 17.00] | 8.50 [0.10 to 18.00] | 4.51 [0.10 to 18.00]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 0 | 98 | 95 | 207
  Male | 9 | 12 | 2 | 89 | 93 | 205
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 25 | 15 | 43
  Not Hispanic or Latino | 9 | 10 | 1 | 134 | 125 | 279
  Unknown or Not Reported | 6 | 7 | 1 | 28 | 48 | 90
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 0 | 3 | 2 | 8
  Asian | 3 | 4 | 0 | 57 | 45 | 109
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 4 | 1 | 23 | 25 | 56
  White | 9 | 7 | 0 | 87 | 93 | 196
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 1 | 17 | 23 | 43

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Pharmacokinetics of LCZ696 Analytes (Sacubitril, LBQ657, and Valsartan): Maximum Drug Concentration in Plasma (Cmax)
Description: The analyses of Cmax was based on plasma concentrations of three sacubitril/valsartan analytes (AHU377 (sacubitril), LBQ657 (sacubitrilat), and valsartan). The plasma levels of sacubitril/valsartan analytes were determined using a validated LCMS/MS method with a lower limit of quantitation (LLOQ) of 1 ng/mL for sacubitril, 20 ng/mL for LBQ657, and 10 ng/mL for valsartan. The PK parameters were determined using the non-compartmental method(s).
Time Frame: Age group 1: Pre-dose and 0.5, 1, 2, 4, 8, 10, optional 24 hours post-dose on Day 1 of Period 1 and 2; Age groups 2 and 3: Pre-dose and 1, 2, 4, 10, optional 24 hours post-dose on Day 1 of Period 1 and 2
Population: Part 1 Pharmacokinetic (PK) Set: included all participants who completed Part 1 screening phase; who had received at least one dose of study drug during Part 1, and had at least one available, valid, PK concentration measurement (not flagged for exclusion or considered a protocol deviation from relevant PK data) during Part 1.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/ml)
Groups:
- LCZ696: 0.8 mg/kg (Age Group 1): Participants received LCZ696 0.8 mg/kg, given as a single oral dose on Day 1 of Period 1 in Part 1. Participants ranging from the age of 6 to less than 18 years were included in this group.
- LCZ696: 0.8 mg/kg (Age Group 2): Participants received LCZ696 0.8 mg/kg, given as a single oral dose on Day 1 of Period 1 in Part 1. Participants ranging from age of 1 to less than 6 years were included in this group.
- LCZ696: 3.1 mg/kg (Age Group 1): Participants received LCZ696 3.1 mg/kg, given as a single oral dose on Day 1 of Period 2 in Part 1. Participants ranging from the age of 6 to less than 18 years were included in this group.
- LCZ696: 3.1 mg/kg (Age Group 2): Participants received LCZ696 3.1 mg/kg, given as a single oral dose on Day 1 of Period 2 in Part 1. Participants ranging from age of 1 to less than 6 years were included in this group.
- LCZ696: 0.4 mg/kg (Age Group 3): Participants received LCZ696 0.4 mg/kg, given as a single oral dose on Day 1 of Period 1 in Part 1. Participants ranging from the age of 1 month to less than 1 year were included in this group.
- LCZ696: 1.6 mg/kg (Age Group 3): Participants received LCZ696 1.6 mg/kg, given as a single oral dose on Day 1 of Period 2 in Part 1. Participants ranging from age 1 month to 1 year were included in this group.
Arm/Group | LCZ696: 0.8 mg/kg (Age Group 1) | LCZ696: 0.8 mg/kg (Age Group 2) | LCZ696: 3.1 mg/kg (Age Group 1) | LCZ696: 3.1 mg/kg (Age Group 2) | LCZ696: 0.4 mg/kg (Age Group 3) | LCZ696: 1.6 mg/kg (Age Group 3)
Number analyzed (Participants) | 7 | 8 | 7 | 6 | 4 | 5
nanograms per milliliter (ng/ml)
  Sacubitril | 523 (390) | 179 (97) | 1970 (1666) | 549 (298) | 124 (80) | 433 (181)
  LBQ657 | 1951 (839) | 1359 (711) | 6707 (1887) | 5453 (1032) | 632 (89) | 2326 (629)
  Valsartan | 1271 (1011) | 1112 (583) | 4035 (1678) | 4935 (1268) | 440 (275) | 2487 (1564)

2. Primary Outcome: Part 1: Pharmacokinetics of LCZ696 Analytes (Sacubitril, LBQ657, and Valsartan): Time to Maximum Plasma Concentration (Tmax)
Description: The analyses of Tmax was based on plasma concentrations of three sacubitril/valsartan analytes (AHU377 (sacubitril), LBQ657 (sacubitrilat), and valsartan). The plasma levels of sacubitril/valsartan analytes were determined using a validated LCMS/MS method with a lower limit of quantitation (LLOQ) of 1 ng/mL for sacubitril, 20 ng/mL for LBQ657, and 10 ng/mL for valsartan. The PK parameters were determined using the non-compartmental method(s).
Time Frame: as for outcome 1
Population: Participants in the Part 1 PK Set were analyzed.
Measure: Mean (Standard Deviation); unit: hours (hr)
Arm/Group | LCZ696: 0.8 mg/kg (Age Group 1) | LCZ696: 0.8 mg/kg (Age Group 2) | LCZ696: 3.1 mg/kg (Age Group 1) | LCZ696: 3.1 mg/kg (Age Group 2) | LCZ696: 0.4 mg/kg (Age Group 3) | LCZ696: 1.6 mg/kg (Age Group 3)
Number analyzed (Participants) | 7 | 8 | 7 | 6 | 4 | 5
hours (hr)
  Sacubitril | 1.1 (1.3) | 1.2 (0.5) | 0.8 (0.3) | 1.2 (0.4) | 1.1 (0.1) | 1.0 (0.0)
  LBQ657 | 4.0 (2.0) | 2.9 (1.1) | 2.9 (1.1) | 3.6 (3.2) | 2.8 (1.6) | 3.6 (0.9)
  Valsartan | 1.7 (1.1) | 2.1 (1.4) | 2.6 (1.0) | 1.9 (0.4) | 1.8 (1.5) | 1.8 (1.3)

3. Primary Outcome: Part 1: Pharmacokinetics of LCZ696 Analytes (Sacubitril, LBQ657, and Valsartan): Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUCinf)
Description: The analyses of AUCinf was based on plasma concentrations of three sacubitril/valsartan analytes (AHU377 (sacubitril), LBQ657 (sacubitrilat), and valsartan). The plasma levels of sacubitril/valsartan analytes were determined using a validated LCMS/MS method with a lower limit of quantitation (LLOQ) of 1 ng/mL for sacubitril, 20 ng/mL for LBQ657, and 10 ng/mL for valsartan. The PK parameters were determined using the non-compartmental method(s).
Time Frame: as for outcome 1
Population: Participants in the Part 1 PK Set were analyzed.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | LCZ696: 0.8 mg/kg (Age Group 1) | LCZ696: 0.8 mg/kg (Age Group 2) | LCZ696: 3.1 mg/kg (Age Group 1) | LCZ696: 3.1 mg/kg (Age Group 2) | LCZ696: 0.4 mg/kg (Age Group 3) | LCZ696: 1.6 mg/kg (Age Group 3)
Number analyzed (Participants) | 7 | 8 | 7 | 6 | 4 | 5
hr*ng/mL
  Sacubitril | 690 (410) | 494 (286) | 3021 (1814) | 1214 (684) | 270 (182) | 1063 (266)
  LBQ657 | 48264 (22939) | 31042 (17259) | 150440 (49515) | 127625 (35634) | 15835 (2912) | 62377 (16035)
  Valsartan | 13540 (12962) | 11036 (7031) | 40733 (21003) | 48561 (21163) | 3923 (1424) | 26170 (16826)

4. Primary Outcome: Part 1: Pharmacokinetics of LCZ696 Analytes (Sacubitril, LBQ657, and Valsartan): Number of Participants With Area Under the Plasma Concentration-time Curve From Time Zero to Last (AUClast)
Description: As prespecified in protocol and SAP the analysis of this outcome measure was done based on dose of LCZ696 administered within the different age groups.
Time Frame: as for outcome 1
Population: Participants in the Part 1 PK Set were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | LCZ696: 0.8 mg/kg (Age Group 1) | LCZ696: 0.8 mg/kg (Age Group 2) | LCZ696: 3.1 mg/kg (Age Group 1) | LCZ696: 3.1 mg/kg (Age Group 2) | LCZ696: 0.4 mg/kg (Age Group 3) | LCZ696: 1.6 mg/kg (Age Group 3)
Number analyzed (Participants) | 7 | 8 | 7 | 6 | 4 | 5
Participants | 7 | 8 | 7 | 6 | 4 | 5

5. Primary Outcome: Part 1: Pharmacokinetics of LCZ696 Analytes (Sacubitril, and Valsartan): Clearance From Plasma (CL/F)
Description: The analyses was based on plasma concentrations of two sacubitril/valsartan analytes (AHU377 (sacubitril), and valsartan). The plasma levels of sacubitril/valsartan analytes were determined using a validated LCMS/MS method with a lower limit of quantitation (LLOQ) of 1 ng/mL for sacubitril, 20 ng/mL for LBQ657, and 10 ng/mL for valsartan. The PK parameters were determined using the non-compartmental method(s). CL/F was not estimated for LBQ657 as it is a metabolite.
Time Frame: as for outcome 1
Population: Participants in the Part 1 PK Set were analyzed.
Measure: Mean (Standard Deviation); unit: liter per hour per kilograms (L/hr/kg)
Arm/Group | LCZ696: 0.8 mg/kg (Age Group 1) | LCZ696: 0.8 mg/kg (Age Group 2) | LCZ696: 3.1 mg/kg (Age Group 1) | LCZ696: 3.1 mg/kg (Age Group 2) | LCZ696: 0.4 mg/kg (Age Group 3) | LCZ696: 1.6 mg/kg (Age Group 3)
Number analyzed (Participants) | 7 | 8 | 7 | 6 | 4 | 5
liter per hour per kilograms (L/hr/kg)
  Sacubitril | 0.73 (0.35) | 1.19 (0.96) | 0.63 (0.28) | 1.67 (1.01) | 1.19 (1.11) | 1.67 (1.01)
  Valsartan | 0.06 (0.05) | 0.07 (0.09) | 0.06 (0.06) | 0.04 (0.01) | 0.06 (0.02) | 0.05 (0.03)

6. Primary Outcome: Part 1: Pharmacokinetics of LCZ696 Analytes (Sacubitril): Time Required to Drug Concentration to Decrease by Half (T 1/2)
Description: The analyses of T1/2 was based on plasma concentrations of sacubitril. The plasma levels of sacubitril/valsartan analytes were determined using a validated LCMS/MS method with a lower limit of quantitation (LLOQ) of 1 ng/mL for sacubitril, 20 ng/mL for LBQ657, and 10 ng/mL for valsartan. The PK parameters were determined using the non-compartmental method(s). T1/2 for other analytes of LCZ696 (LBQ657 and Valsartan) was not estimable due to the short sample collection timeframe.
Time Frame: as for outcome 1
Population: Part 1 PK Set. The overall number of participants analyzed is the number of participants with data available for this endpoint. T1/2 could not be determined for participants under the arm LCZ696: 0.4 mg/kg (Age Group 3) as their PK data was inadequate for the T1/2 calculation. As participants were from the age of 1 month to less than 1 year, it was difficult to obtain multiple PK samples.
Measure: Median (Full Range); unit: hours
Arm/Group | LCZ696: 0.8 mg/kg (Age Group 1) | LCZ696: 0.8 mg/kg (Age Group 2) | LCZ696: 3.1 mg/kg (Age Group 1) | LCZ696: 3.1 mg/kg (Age Group 2) | LCZ696: 0.4 mg/kg (Age Group 3) | LCZ696: 1.6 mg/kg (Age Group 3)
Number analyzed (Participants) | 6 | 2 | 6 | 4 | 0 | 3
hours | 1.26 [0.95 to 2.36] | 1.53 [1.40 to 1.65] | 1.34 [1.16 to 1.60] | 1.51 [1.34 to 1.70] |  | 1.33 [1.16 to 1.64]

7. Primary Outcome: Part 1: Pharmacodynamics (PD) of LCZ696 Analytes (Sacubitril, LBQ657, and Valsartan): Change From Baseline in Plasma B-type Natriuretic Peptide (BNP)
Description: Biomarkers were used to assess the PD effects of LCZ696. Blood biomarkers of potential interest included plasma BNP. Biomarkers related to heart failure or the mechanism of action of the study drug were measured. Summary statistics for change from baseline at each time point is presented. The baseline assessment is defined as the last non-missing assessment (scheduled or unscheduled) prior to (the first dose time of the study drug within the dose associated period). For each post-dose time point, participants are included if and only if the participant has both pre-dose assessment and current time point assessment observed.
Time Frame: Baseline (0 hrs pre dose), 4 and 8 hrs post dose on Day 1 of Period 1 and Period 2
Population: Part 1 PD set (PD1) included all participants who completed the Part 1 screening phase and had at least one dose of study drug during Part 1 of the study, at least one available PD measurement during Part 1 of the study and with no protocol deviations with relevant impact on PD data. Overall number of participants analyzed is the number of participants with data available for this endpoint.
Measure: Geometric Mean (95% Confidence Interval); unit: picomoles per liter (pmol/L)
Arm/Group | LCZ696: 0.8 mg/kg (Age Group 1) | LCZ696: 0.8 mg/kg (Age Group 2) | LCZ696: 3.1 mg/kg (Age Group 1) | LCZ696: 3.1 mg/kg (Age Group 2) | LCZ696: 0.4 mg/kg (Age Group 3) | LCZ696: 1.6 mg/kg (Age Group 3)
Number analyzed (Participants) | 6 | 6 | 7 | 3 | 3 | 4
picomoles per liter (pmol/L)
  Baseline (0 hrs pre dose) | 100.87 [49.84 to 204.13] | 63.80 [8.65 to 470.81] | 97.52 [51.59 to 184.32] | 120.51 [5.21 to 2787.44] | 21.20 [2.14 to 210.41] | 129.29 [9.45 to 1768.43]
  Change From Baseline (4 hrs post dose): number analyzed (Participants) | 6 | 4 | 7 | 1 | 3 | 4
  Change From Baseline (4 hrs post dose) | 1.31 [0.93 to 1.85] | 1.60 [0.21 to 11.95] | 1.22 [0.94 to 1.58] | 0.62 [NA to NA] — The 95% confidence interval (CI) was not estimable for one participant | 0.77 [0.56 to 1.05] | 1.09 [0.61 to 1.93]
  Change From Baseline (8 hrs post dose): number analyzed (Participants) | 5 | 4 | 1 | 1 | 3 | 2
  Change From Baseline (8 hrs post dose) | 1.32 [0.92 to 1.88] | 1.21 [0.21 to 7.04] | 0.97 [0.70 to 1.34] | 0.80 [NA to NA] — The 95% CI was not estimable for one participant | 0.59 [0.27 to 1.30] | 0.55 [0.15 to 2.02]

8. Primary Outcome: Part 1: Pharmacodynamics of LCZ696 Analytes (Sacubitril, LBQ657, and Valsartan): Change From Baseline in Plasma N-terminal Pro-brain Natriuretic Peptide (NTproBNP)
Description: Biomarkers were used to assess the PD effects of LCZ696. Blood biomarkers of potential interest included plasma NTproBNP. Biomarkers related to heart failure or the mechanism of action of the study drug were measured. Summary statistics for change from baseline at each time point is presented. The baseline assessment is defined as the last non-missing assessment (scheduled or unscheduled) prior to (the first dose time of the study drug within the dose associated period). For each post-dose time point, participants are included if and only if the participant has both pre-dose assessment and current time point assessment observed.
Time Frame: Baseline (0 hrs pre dose) and optional 24 hrs post dosing on Day 1 of Period 1 and Period 2
Population: Part 1 PD set. The overall number of participants analyzed is the number of participants with data available for this endpoint. Data has not been reported for the arms of LCZ696: 0.8 mg/kg (Age Group 2) and LCZ696: 3.1 mg/kg (Age Group 2) as no participants participated in the optional 24 hrs post-dose assessment.
Measure: Geometric Mean (95% Confidence Interval); unit: picograms per millilitre (pg/mL)
Arm/Group | LCZ696: 0.8 mg/kg (Age Group 1) | LCZ696: 0.8 mg/kg (Age Group 2) | LCZ696: 3.1 mg/kg (Age Group 1) | LCZ696: 3.1 mg/kg (Age Group 2) | LCZ696: 0.4 mg/kg (Age Group 3) | LCZ696: 1.6 mg/kg (Age Group 3)
Number analyzed (Participants) | 7 | 0 | 7 | 0 | 4 | 5
picograms per millilitre (pg/mL)
  Baseline (0 hrs pre dose) | 2385.34 [1186.13 to 4796.98] |  | 2179.94 [932.77 to 5094.69] |  | 961.76 [125.65 to 7361.70] | 5086.37 [683.53 to 37849.47]
  Change From Baseline (24 hrs post dose): number analyzed (Participants) | 3 | 0 | 0 | 0 | 2 | 2
  Change From Baseline (24 hrs post dose) | 0.74 [0.31 to 1.78] |  |  |  | 0.59 [0.00 to 134.25] | 0.41 [0.34 to 0.48]

9. Primary Outcome: Part 1: Pharmacodynamics of LCZ696 Analytes (Sacubitril, LBQ657, and Valsartan): Change From Baseline in Plasma Cyclic Guanosine Monophosphate (cGMP)
Description: Biomarkers were used to assess the PD effects of LCZ696. Blood biomarkers of potential interest included plasma cGMP. Biomarkers related to heart failure or the mechanism of action of the study drug were measured. Summary statistics for change from baseline at each time point is presented. The baseline assessment is defined as the last non-missing assessment (scheduled or unscheduled) prior to (the first dose time of the study drug within the dose associated period). For each post-dose time point, participants are included if and only if the participant has both pre-dose assessment and current time point assessment observed.
Time Frame: Baseline (0 hrs pre dose), 4 and 8 hrs post dose on Day 1 of Period 1 and Period 2
Population: Part 1 PD set. The overall number of participants analyzed is the number of participants with data available for this endpoint.
Measure: Geometric Mean (95% Confidence Interval); unit: nanomoles per litre (nmol/L)
Arm/Group | LCZ696: 0.8 mg/kg (Age Group 1) | LCZ696: 0.8 mg/kg (Age Group 2) | LCZ696: 3.1 mg/kg (Age Group 1) | LCZ696: 3.1 mg/kg (Age Group 2) | LCZ696: 0.4 mg/kg (Age Group 3) | LCZ696: 1.6 mg/kg (Age Group 3)
Number analyzed (Participants) | 7 | 6 | 7 | 4 | 2 | 3
nanomoles per litre (nmol/L)
  Baseline (0 hrs pre dose) | 18.18 [12.01 to 27.51] | 21.41 [12.83 to 35.71] | 12.20 [8.13 to 18.32] | 24.55 [18.37 to 32.82] | 13.38 [0.05 to 3883.59] | 22.84 [12.51 to 41.68]
  Change From Baseline (4 hrs post dose) | 1.30 [0.89 to 1.90] | 0.90 [0.50 to 1.62] | 1.54 [1.12 to 2.10] | 1.02 [0.52 to 2.01] | 0.80 [0.00 to 618.02] | 0.78 [0.27 to 2.22]
  Change From Baseline (8 hrs post dose): number analyzed (Participants) | 7 | 4 | 7 | 4 | 2 | 3
  Change From Baseline (8 hrs post dose) | 1.17 [0.91 to 1.50] | 0.92 [0.66 to 1.29] | 1.60 [1.10 to 2.31] | 0.40 [0.02 to 8.86] | 0.79 [0.00 to 230.10] | 0.79 [0.29 to 2.18]

10. Primary Outcome: Part 1: Pharmacodynamics of LCZ696 Analytes (Sacubitril, LBQ657, and Valsartan): Change From Baseline in Urine cGMP
Description: Biomarkers were used to assess the PD effects of LCZ696. Blood biomarkers of potential interest included urine cGMP. Biomarkers related to heart failure or the mechanism of action of the study drug were measured. Summary statistics for change from baseline at each time point is presented. The baseline assessment is defined as the last non-missing assessment (scheduled or unscheduled) prior to (the first dose time of the study drug within the dose associated period). For each post-dose time point, participants are included if and only if the participant has both pre-dose assessment and current time point assessment observed.
Time Frame: Baseline (0 hrs pre dose), 4 to 8 hrs post dose on Day 1 of Period 1 and Period 2
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | LCZ696: 0.8 mg/kg (Age Group 1) | LCZ696: 0.8 mg/kg (Age Group 2) | LCZ696: 3.1 mg/kg (Age Group 1) | LCZ696: 3.1 mg/kg (Age Group 2) | LCZ696: 0.4 mg/kg (Age Group 3) | LCZ696: 1.6 mg/kg (Age Group 3)
Number analyzed (Participants) | 7 | 3 | 6 | 3 | 2 | 5
nmol/L
  Baseline (0 hrs pre dose): number analyzed (Participants) | 7 | 3 | 6 | 3 | 1 | 5
  Baseline (0 hrs pre dose) | 1055.56 [352.98 to 3156.55] | 1349.91 [118.48 to 15380.33] | 914.57 [311.65 to 2683.88] | 1123.69 [75.21 to 16789.03] | 485.00 [NA to NA] — The 95% CI was not estimable for one participant | 386.32 [134.04 to 1113.42]
  Change From Baseline (4 to 8 hrs post dose): number analyzed (Participants) | 7 | 3 | 6 | 3 | 2 | 4
  Change From Baseline (4 to 8 hrs post dose) | 1.42 [0.38 to 5.32] | 0.80 [0.02 to 27.03] | 1.79 [0.65 to 4.96] | 2.17 [0.10 to 45.16] | 0.92 [0.02 to 51.75] | 1.98 [0.51 to 7.63]

11. Primary Outcome: Part 2: Percentage of Participants With Worst Event in Each Category Based on Global Ranking
Description: Global ranking is based on 5 categories ranking worst to best outcome:Category 1:Death; United Network for Organ Sharing(UNOS)status 1A listing for heart transplant or equivalent; ventricular assist device(VAD)/extracorporeal membrane oxygenation(ECMO)/mechanical ventilation/intra-aortic balloon pump requirement for life support at end of study. Category 2:Worsening HF(WHF);defined by signs and symptoms of WHF that requires an intensification of HF therapy. Category 3:Worsened; worse New York Heart Association(NYHA)/Ross or worse Patient Global Impression of Severity(PGIS); and further ranking by Pediatric Quality of Life Inventory(PedsQL)physical functioning domain.Category 4:Unchanged; unchanged NYHA/Ross and unchanged PGIS; and further ranking by PedsQL physical functioning domain. Category 5:Improved; improved NYHA/Ross or improved PGIS(neither can be worse);and further ranking by PedsQL physical functioning domain. Participants with worst event in each category are reported here.
Time Frame: Up to 52 weeks
Population: Full analysis set included all randomized participants with the exception of those participants who had not been qualified for randomization and had not received study drug but had been inadvertently randomized into the study. A total of 377 participants were randomized in Part 2 of which a total of 375 were analyzed. Two participants who were excluded did not receive study drug and did not qualify for randomization.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: LCZ696 | Part 2: Enalapril
Number analyzed (Participants) | 187 | 188
percentage of participants
  Category 1 | 10.16 | 15.96
  Category 2 | 9.63 | 4.79
  Category 3 | 6.95 | 5.85
  Category 4 | 20.86 | 26.60
  Category 5 | 39.57 | 35.64
  Missing | 12.83 | 11.17

12. Secondary Outcome: Part 1: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence associated with use of a drug in humans, whether considered drug related or not, that occurs after a participant provides informed consent. TEAEs during part 1 are defined as any recorded AE with its start date (recorded or imputed) later than or equal to the date of the first dose of the study drug within part 1 and its start date prior to or equal to the end date of the part 1.
Time Frame: From first dose to 30 days after last dose of study drug in Part 1
Population: Part 1 Safety Analysis Set (SAF1) included all participants who completed the Part 1 screening phase and received at least one dose of study drug during Part 1 of the study.
Measure: Number; unit: percentage of participants
Groups:
- LCZ696: 0.8 mg/kg (Age Group 1): Participants received LCZ696 0.4 mg/kg (age group 3 {1 month to < 1 year}) or 0.8 mg/kg (age group 1 {6 to <18 years} and age group 2 {1 to < 6 years}), based on age, given as a single oral dose on Day 1 of period 1.
Arm/Group | LCZ696: 0.8 mg/kg (Age Group 1) | LCZ696: 0.8 mg/kg (Age Group 2) | LCZ696: 3.1 mg/kg (Age Group 1) | LCZ696: 3.1 mg/kg (Age Group 2) | LCZ696: 0.4 mg/kg (Age Group 3) | LCZ696: 1.6 mg/kg (Age Group 3) | Part 1: Dose Cohort S
Number analyzed (Participants) | 7 | 6 | 7 | 6 | 4 | 5 | 2
percentage of participants | 28.57 | 50.00 | 28.57 | 50.00 | 50.00 | 80.00 | 50.00

13. Secondary Outcome: Part 2: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An AE is any untoward medical occurrence associated with use of a drug in humans, whether or not considered drug related, that occurs after a participant provides informed consent. TEAEs during part 2 are defined as any recorded AE with its start date (recorded or imputed) later than or equal to the date of the first dose of the study drug within part 2 and its start date prior to or equal to the end date of part 2.
Time Frame: From first dose to 30 days after last dose of study drug in Part 2 (up to 56 weeks)
Population: Part 2: Safety Set included randomized participants who received at least one dose of study drug. Participants were analyzed according to the treatment actually received. A total of 377 participants were randomized in Part 2 of which a total of 375 were analyzed. Two participants who were excluded did not receive study drug and did not qualify for randomization.
Measure: Number; unit: percentage of participant
Arm/Group | Part 2: LCZ696 | Part 2: Enalapril
Number analyzed (Participants) | 187 | 188
percentage of participant | 88.77 | 87.77

14. Secondary Outcome: Part 2: Exposure-adjusted Incidence Rate of Category 1 or Category 2 Event
Description: The exposure adjusted incidence rate is calculated as number of participants with at least one event divided by total participant years across all participants. Category 1: Death; UNOS status 1A listing for heart transplant or equivalent; VAD/ECMO/mechanical ventilation/intra-aortic balloon pump requirement for life support at end of study. Category 2: WHF; defined by signs and symptoms of WHF that requires an intensification of HF therapy.
Time Frame: 52 weeks
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: participant per participant years
Arm/Group | Part 2: LCZ696 | Part 2: Enalapril
Number analyzed (Participants) | 34 | 33
participant per participant years | 20.133 [13.9430 to 28.1344] | 20.042 [13.7960 to 28.1464]
Statistical Analysis 1: Comparison: Part 2: LCZ696 vs Part 2: Enalapril; Test type: Superiority; p = 0.7958, Cox Proportional Hazard — The adjusted hazard ratio and the p-values are based on a Cox proportional hazard model, stratified by modified age group with treatment and NYHA/ROSS class group included as factor; Cox Proportional Hazard = 1.0655, 95% CI 2-sided [0.6589 to 1.7232]

15. Secondary Outcome: Part 2: Percentage of Participants With Change From Baseline in New York Heart Association (NYHA)/Ross Functional Class
Description: NYHA classification is a subjective physician's assessment of participant's functional capacity and symptomatic status and can change frequently over time. NYHA is tool that classifies participants with heart failure into one of four classes according to their degree of symptoms at rest and with activity. Class I: No limitations of physical activity. Class 2: May experience fatigue, palpitations, dyspnea, or angina during moderate exercise but not during rest. Class 3: Symptoms with minimal exertion that interfere with normal daily activity. Class 4: Unable to carry out any physical activity because they typically have symptoms of HF at rest that worsen with any exertion. Participants with change from baseline were classified as improved (shifted from higher to lower class), unchanged (no change in class) or worsened (shifted from lower to higher class).
Time Frame: Baseline, Week 4, 12, 24, 36, and 52
Population: Participants in the full analysis set with available data were analyzed. The number analyzed is the number of participants with data available for analyses at specific timepoints. A total of 377 participants were randomized in Part 2 of which a total of 375 were analyzed. Two participants who were excluded did not receive study drug and did not qualify for randomization.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: LCZ696 | Part 2: Enalapril
Number analyzed (Participants) | 187 | 188
percentage of participants
  Change from Baseline at Week 4: Improved: number analyzed (Participants) | 183 | 184
  Change from Baseline at Week 4: Improved | 14.21 | 15.67
  Change from Baseline at Week 4: Unchanged: number analyzed (Participants) | 183 | 184
  Change from Baseline at Week 4: Unchanged | 84.15 | 82.61
  Change from Baseline at Week 4: Worsened: number analyzed (Participants) | 183 | 184
  Change from Baseline at Week 4: Worsened | 1.64 | 1.63
  Change from Baseline at Week 12: Improved: number analyzed (Participants) | 180 | 180
  Change from Baseline at Week 12: Improved | 23.89 | 25.56
  Change from Baseline at Week 12: Unchanged: number analyzed (Participants) | 180 | 180
  Change from Baseline at Week 12: Unchanged | 70.56 | 67.78
  Change from Baseline at Week 12: Worsened: number analyzed (Participants) | 180 | 180
  Change from Baseline at Week 12: Worsened | 5.56 | 6.67
  Change from Baseline at Week 24: Improved: number analyzed (Participants) | 178 | 172
  Change from Baseline at Week 24: Improved | 26.97 | 27.91
  Change from Baseline at Week 24: Unchanged: number analyzed (Participants) | 178 | 172
  Change from Baseline at Week 24: Unchanged | 64.04 | 63.95
  Change from Baseline at Week 24: Worsened: number analyzed (Participants) | 178 | 172
  Change from Baseline at Week 24: Worsened | 8.99 | 8.14
  Change from Baseline at Week 36: Improved: number analyzed (Participants) | 167 | 170
  Change from Baseline at Week 36: Improved | 29.94 | 34.12
  Change from Baseline at Week 36: Unchanged: number analyzed (Participants) | 167 | 170
  Change from Baseline at Week 36: Unchanged | 61.08 | 58.24
  Change from Baseline at Week 36: Worsened: number analyzed (Participants) | 167 | 170
  Change from Baseline at Week 36: Worsened | 8.98 | 7.65
  Change from Baseline at Week 52: Improved: number analyzed (Participants) | 154 | 159
  Change from Baseline at Week 52: Improved | 37.66 | 33.96
  Change from Baseline at Week 52: Unchanged: number analyzed (Participants) | 154 | 159
  Change from Baseline at Week 52: Unchanged | 50.65 | 56.60
  Change from Baseline at Week 52: Worsened: number analyzed (Participants) | 154 | 159
  Change from Baseline at Week 52: Worsened | 11.69 | 9.43

16. Secondary Outcome: Part 2: Percentage of Participants With Change From Baseline in Patient Global Impression of Severity (PGIS) Score
Description: PGIS of Heart Failure Symptoms is a 1-item questionnaire to assess the participant's impression of symptoms severity, specifically: shortness of breath, fatigue and swelling. The PGI-S asks the participant to choose one response that best describes how his/her heart failure symptoms, specifically: shortness of breath, fatigue and swelling are now on a 5-point scale, ranging from 'Not at all' (1) to 'Very severe' (5). C1 = none (good), C2 = mild, C3 = moderate, C4 = severe, C5 = very severe (bad). Percentage of participants by change in score are reported. Participants with change from baseline were classified as improved (shifted from higher to score), unchanged (no change in score) or worsened (shifted from lower to higher score).
Time Frame: Baseline, Week 4, 12, 24, 36, and 52
Population: Participants in the full analysis set with available data were analyzed. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analyses at specific timepoints. A total of 377 participants were randomized in Part 2 of which a total of 375 were analyzed. Two participants who were excluded did not receive study drug and did not qualify for randomization.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2: LCZ696 | Part 2: Enalapril
Number analyzed (Participants) | 182 | 188
percentage of participants
  Change from Baseline at Week 4: Improved: number analyzed (Participants) | 174 | 182
  Change from Baseline at Week 4: Improved | 27.01 | 29.67
  Change from Baseline at Week 4: Unchanged: number analyzed (Participants) | 174 | 182
  Change from Baseline at Week 4: Unchanged | 58.05 | 59.89
  Change from Baseline at Week 4: Worsened: number analyzed (Participants) | 174 | 182
  Change from Baseline at Week 4: Worsened | 14.94 | 10.44
  Change from Baseline at Week 12: Improved: number analyzed (Participants) | 178 | 178
  Change from Baseline at Week 12: Improved | 30.90 | 31.46
  Change from Baseline at Week 12: Unchanged: number analyzed (Participants) | 178 | 178
  Change from Baseline at Week 12: Unchanged | 52.25 | 55.62
  Change from Baseline at Week 12: Worsened: number analyzed (Participants) | 178 | 178
  Change from Baseline at Week 12: Worsened | 16.85 | 12.92
  Change from Baseline at Week 24: Improved: number analyzed (Participants) | 174 | 171
  Change from Baseline at Week 24: Improved | 33.33 | 38.01
  Change from Baseline at Week 24: Unchanged: number analyzed (Participants) | 174 | 171
  Change from Baseline at Week 24: Unchanged | 48.85 | 48.54
  Change from Baseline at Week 24: Worsened: number analyzed (Participants) | 174 | 171
  Change from Baseline at Week 24: Worsened | 17.82 | 13.45
  Change from Baseline at Week 36: Improved: number analyzed (Participants) | 162 | 165
  Change from Baseline at Week 36: Improved | 33.33 | 33.94
  Change from Baseline at Week 36: Unchanged: number analyzed (Participants) | 162 | 165
  Change from Baseline at Week 36: Unchanged | 49.38 | 52.73
  Change from Baseline at Week 36: Worsened: number analyzed (Participants) | 162 | 165
  Change from Baseline at Week 36: Worsened | 17.28 | 13.33
  Change from Baseline at Week 52: Improved: number analyzed (Participants) | 152 | 158
  Change from Baseline at Week 52: Improved | 35.53 | 34.81
  Change from Baseline at Week 52: Unchanged: number analyzed (Participants) | 152 | 158
  Change from Baseline at Week 52: Unchanged | 48.03 | 47.47
  Change from Baseline at Week 52: Worsened: number analyzed (Participants) | 152 | 158
  Change from Baseline at Week 52: Worsened | 16.45 | 17.72

17. Secondary Outcome: Part 1 and Part 2: Population PK of LCZ696 Analytes: Clearance From Plasma (CL)
Description: The analyses of CL was based on plasma concentrations of three sacubitril/valsartan analytes (AHU377 (sacubitril), LBQ657 (sacubitrilat), and valsartan). The PK parameters were determined using the non-compartmental method(s). In case of data limitations for estimating PK parameters using non-compartmental methods, a population PK approach was used to estimate exposure of sacubitril/valsartan analytes. The population PK model was developed to describe incoming data from pediatric patients based on an established model developed for the adult population.
Time Frame: Part 1: Age group 1- Pre-dose and 0.5, 1, 2, 4, 8, 10, optional 24 hours post-dose on Day 1 of Period 1 and 2; Age groups 2 and 3- Pre-dose and 1, 2, 4, 10, optional 24 hours post-dose on Day 1 of Period 1 and 2; Part 2: Weeks 2, 8, 12, 52
Population: The Full Analysis Set included all randomized participants who received study drug, with the exception of [2 patients in Part 2] who had not received any study drug but had been inadvertently randomized into the study (mis-randomized).
Measure: Mean (Standard Deviation); unit: L/h
Groups:
- LCZ696 (Part 1 and 2): Participants received LCZ696 0.4 mg/kg (age group 3) or 0.8 mg/kg (age group 1 and 2) on Day 1 of Period 1 and 1.6 mg/kg (age group 3) or 3.1 mg/kg (age group 1 and 2) on Day 1 of Period 2, based on age, given as a single oral dose in Part 1. Followed by Part 1, participants were enrolled in Part 2 and received LCZ696 2.3 mg/kg (age group 3) or 3.1 mg/kg (age group 1 and 2), based on age, orally, twice a day (BID) for 52 weeks in Part 2.
Arm/Group | LCZ696 (Part 1 and 2)
Number analyzed (Participants) | 203
L/h
  Sacubitril: number analyzed (Participants) | 202
  Sacubitril | 25.93 (19.29)
  LBQ657: number analyzed (Participants) | 202
  LBQ657 | 0.44 (0.31)
  Valsartan | 1.97 (1.69)

18. Secondary Outcome: Part 1 and Part 2: Population PK of LCZ696 Analytes: Volume of Distribution in Steady State
Description: The analyses of volume of distribution was based on plasma concentrations of three sacubitril/valsartan analytes (AHU377 (sacubitril), LBQ657 (sacubitrilat), and valsartan). The PK parameters were determined using the non-compartmental method(s). In case of data limitations for estimating PK parameters using non-compartmental methods, a population PK approach was used to estimate exposure of sacubitril/valsartan analytes. The population PK model was developed to describe incoming data from pediatric patients based on an established model developed for the adult population.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: L/Kg
Arm/Group | LCZ696 (Part 1 and 2)
Number analyzed (Participants) | 203
L/Kg
  Sacubitril: number analyzed (Participants) | 202
  Sacubitril | 4.67 (5.84)
  LBQ657: number analyzed (Participants) | 202
  LBQ657 | 0.34 (0.12)
  Valsartan | 0.68 (0.29)

19. Secondary Outcome: Part 1 and Part 2: Population PK of LCZ696 Analytes: Absorption Rate Constant (Ka)
Description: The analyses of Ka was based on plasma concentrations of three sacubitril/valsartan analytes (AHU377 (sacubitril), LBQ657 (sacubitrilat), and valsartan). The PK parameters were determined using the non-compartmental method(s). In case of data limitations for estimating PK parameters using non-compartmental methods, a population PK approach was used to estimate exposure of sacubitril/valsartan analytes. The population PK model was developed to describe incoming data from pediatric patients based on an established model developed for the adult population.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | LCZ696 (Part 1 and 2)
Number analyzed (Participants) | 203
1/hour
  Sacubitril: number analyzed (Participants) | 202
  Sacubitril | 1.25 (0.01)
  LBQ657: number analyzed (Participants) | 202
  LBQ657 | 1.04 (1.34)
  Valsartan | 1.42 (0.92)

20. Secondary Outcome: Part 1 and Part 2: Population PK of LCZ696 Analytes: Time Required to Drug Concentration to Decrease by Half (T 1/2)
Description: The analyses of T1/2 was based on plasma concentrations of three sacubitril/valsartan analytes (AHU377 (sacubitril), LBQ657 (sacubitrilat), and valsartan). The PK parameters were determined using the non-compartmental method(s). In case of data limitations for estimating PK parameters using non-compartmental methods, a population PK approach was used to estimate exposure of sacubitril/valsartan analytes. The population PK model was developed to describe incoming data from pediatric patients based on an established model developed for the adult population.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Median (Full Range); unit: hours
Arm/Group | LCZ696 (Part 1 and 2)
Number analyzed (Participants) | 203
hours
  Sacubitril: number analyzed (Participants) | 202
  Sacubitril | 8.51 [1.87 to 199.55]
  LBQ657: number analyzed (Participants) | 202
  LBQ657 | 18.21 [6.08 to 107.47]
  Valsartan | 7.96 [2.33 to 81.65]

21. Secondary Outcome: Part 1 and Part 2: Population PK of LCZ696 Analytes: Maximum Drug Concentration in Plasma at Steady State (Cmax,ss)
Description: The analyses of Cmax was based on plasma concentrations of three sacubitril/valsartan analytes (AHU377 (sacubitril), LBQ657 (sacubitrilat), and valsartan). The PK parameters were determined using the non-compartmental method(s). In case of data limitations for estimating PK parameters using non-compartmental methods, a population PK approach was used to estimate exposure of sacubitril/valsartan analytes. The population PK model was developed to describe incoming data from pediatric patients based on an established model developed for the adult population.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LCZ696 (Part 1 and 2)
Number analyzed (Participants) | 203
ng/mL
  Sacubitril: number analyzed (Participants) | 202
  Sacubitril | 1348 (627)
  LBQ657: number analyzed (Participants) | 202
  LBQ657 | 10153 (3591)
  Valsartan | 3861 (1770)

22. Secondary Outcome: Part 1 and Part 2: Population PK of LCZ696 Analytes: Lowest Plasma Concentration Observed During a Dosing Interval at Steady State (Cmin,ss)
Description: The analyses of Cmin was based on plasma concentrations of three sacubitril/valsartan analytes (AHU377 (sacubitril), LBQ657 (sacubitrilat), and valsartan). The PK parameters were determined using the non-compartmental method(s). In case of data limitations for estimating PK parameters using non-compartmental methods, a population PK approach was used to estimate exposure of sacubitril/valsartan analytes. The population PK model was developed to describe incoming data from pediatric patients based on an established model developed for the adult population.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LCZ696 (Part 1 and 2)
Number analyzed (Participants) | 203
ng/mL
  Sacubitril: number analyzed (Participants) | 202
  Sacubitril | 63 (141)
  LBQ657: number analyzed (Participants) | 202
  LBQ657 | 6442 (3474)
  Valsartan | 1442 (1564)

23. Secondary Outcome: Part 1 and Part 2: Population PK of LCZ696 Analytes: Area Under the Plasma Concentration-time Curve From Time Zero to the End of the Dosing Interval Tau at Steady State (AUCtau,ss)
Description: The analyses of AUCtau was based on plasma concentrations of three sacubitril/valsartan analytes (AHU377 (sacubitril), LBQ657 (sacubitrilat), and valsartan). The PK parameters were determined using the non-compartmental method(s). In case of data limitations for estimating PK parameters using non-compartmental methods, a population PK approach was used to estimate exposure of sacubitril/valsartan analytes. The population PK model was developed to describe incoming data from pediatric patients based on an established model developed for the adult population.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng/mL*h
Arm/Group | LCZ696 (Part 1 and 2)
Number analyzed (Participants) | 203
ng/mL*h
  Sacubitril | 2179 (2241)
  LBQ657 | 98906 (41944)
  Valsartan | 28672 (19686)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment plus 30 days post treatment up to approximately one year.
Description: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment.
  Of the 26 participants enrolled in Part 1, all 26 participants received at least one dose of study medication. Of the 377 participants enrolled in Part 2, 375 received study medication. 2 participants in the Enalapril arm were mis-randomized in error; therefore, did not receive any medication.
Arm/Group | Part 1: Dose Cohort 1 | Part 1: Dose Cohort 2 | Part 1: Dose Cohort S | Part 2: LCZ696 | Part 2: Enalapril
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/18 | 0/2 | 8/187 | 12/188
Serious Adverse Events (participants affected / at risk) | 2/17 | 1/18 | 0/2 | 69/187 | 62/188
Other Adverse Events (participants affected / at risk) | 6/17 | 10/18 | 1/2 | 161/187 | 156/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Dose Cohort 1 (N=17) | Part 1: Dose Cohort 2 (N=18) | Part 1: Dose Cohort S (N=2) | Part 2: LCZ696 (N=187) | Part 2: Enalapril (N=188)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 3
Arrhythmia supraventricular (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Atrial thrombosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 2
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 2 | 4
Cardiac disorder (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 24 | 23
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 0 | 2 | 4
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 4 | 3
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Pulseless electrical activity (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 3 | 1
Adrenogenital syndrome (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Intussusception (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 5 | 4
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 2
Death (General disorders) | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 4 | 0
Sudden death (General disorders) | 0 | 0 | 0 | 1 | 0
Heart transplant rejection (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Bronchitis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 0 | 2 | 2
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 5 | 4
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia mycoplasmal (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 4 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Viral sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 2
Accidental exposure to product (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Anticoagulation drug level above therapeutic (Investigations) | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 1
Cardiac output decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Coronavirus test positive (Investigations) | 0 | 0 | 0 | 1 | 0
Human rhinovirus test positive (Investigations) | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Feeding intolerance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Akinesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Basal ganglia infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Brain injury (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Febrile convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Juvenile myoclonic epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Neuromyopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Partial seizures (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1 | 4
Status epilepticus (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 2
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 2
Renal artery stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 4 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Dose Cohort 1 (N=17) | Part 1: Dose Cohort 2 (N=18) | Part 1: Dose Cohort S (N=2) | Part 2: LCZ696 (N=187) | Part 2: Enalapril (N=188)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 7 | 5
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 3 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 2
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 2 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 5 | 6
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 2 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 2 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 4
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 4
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 2 | 3
Phimosis (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 2 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 15 | 11
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 6 | 9
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 6 | 7
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 25 | 23
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 5 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 9 | 9
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 5 | 2
Vomiting (Gastrointestinal disorders) | 1 | 4 | 1 | 33 | 37
Asthenia (General disorders) | 0 | 0 | 0 | 3 | 2
Chest discomfort (General disorders) | 0 | 0 | 0 | 2 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 7 | 7
Face oedema (General disorders) | 0 | 0 | 0 | 1 | 2
Fatigue (General disorders) | 0 | 1 | 1 | 19 | 14
Medical device pain (General disorders) | 0 | 0 | 0 | 2 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 2 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 7 | 2
Peripheral swelling (General disorders) | 0 | 1 | 1 | 0 | 2
Pyrexia (General disorders) | 0 | 1 | 0 | 36 | 34
Swelling face (General disorders) | 0 | 1 | 1 | 1 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 3 | 2
Acarodermatitis (Infections and infestations) | 0 | 0 | 0 | 0 | 3
Atypical pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 12 | 8
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 6 | 2
Candida infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 2 | 3
Exanthema subitum (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 9 | 11
Gastroenteritis rotavirus (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 3 | 2
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 0 | 0 | 2 | 3
Influenza (Infections and infestations) | 0 | 0 | 0 | 11 | 12
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 29 | 17
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 3
Otitis media (Infections and infestations) | 0 | 0 | 0 | 5 | 3
Otitis media acute (Infections and infestations) | 0 | 0 | 0 | 2 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 6 | 5
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 3 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 3 | 3
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 2 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 4 | 5
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 7 | 10
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 3 | 2
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 3
Tracheitis (Infections and infestations) | 0 | 0 | 0 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 3 | 1 | 37 | 35
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 5 | 4
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 3
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2 | 5
Lip injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 4
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 2
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 2
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 3 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 3 | 1
Blood creatine increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 6 | 5
Blood potassium increased (Investigations) | 0 | 0 | 0 | 3 | 2
Blood urea increased (Investigations) | 1 | 0 | 0 | 2 | 1
Blood uric acid increased (Investigations) | 1 | 1 | 0 | 1 | 2
Body temperature increased (Investigations) | 0 | 1 | 0 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 0 | 9 | 12
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1 | 2
SARS-CoV-2 test negative (Investigations) | 0 | 0 | 0 | 6 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 4
Weight increased (Investigations) | 0 | 0 | 0 | 3 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 9 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 6 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 4 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 4 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 6 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 6 | 3
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 23 | 15
Headache (Nervous system disorders) | 0 | 0 | 0 | 22 | 20
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Migraine (Nervous system disorders) | 0 | 0 | 0 | 2 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 3
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 3 | 5
Depression (Psychiatric disorders) | 0 | 0 | 0 | 2 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 4 | 3
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 3 | 2
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0
Renal failure (Renal and urinary disorders) | 1 | 1 | 0 | 1 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 4 | 2
Balanoposthitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 2
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 36 | 38
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 6 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 9 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 9 | 5
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 5 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 7 | 7
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 4 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 4 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 5 | 6
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 2
Hypotension (Vascular disorders) | 1 | 2 | 0 | 21 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (3):
  • Study Protocol (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/12/NCT02678312/Prot_000.pdf
  • Statistical Analysis Plan: Original Statistical Analysis Plan (SAP) (2021-10-29): https://cdn.clinicaltrials.gov/large-docs/12/NCT02678312/SAP_001.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan (SAP) for China Sub-CSR (2021-10-25): https://cdn.clinicaltrials.gov/large-docs/12/NCT02678312/SAP_002.pdf